CLINICAL TRIAL: NCT07092020
Title: A Prospective, Randomized, Controlled, Observer-masked, Multi-center Clinical Trial to Demonstrate the Safety and Effectiveness of the Extended Depth of Focus AT LARA 829MP Posterior Chamber Intraocular Lens for Correction of Aphakia
Brief Title: EDF IOL Versus Monofocal IOL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AT LARA 829MP BER-401-24
Record Dates: First submitted 2025-07-11; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Cataract Senile
Keywords: IOL; Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EDF (Experimental): Extended depth of focus
  Interventions: Device: EDF
- Monofocal (Active Comparator): Monofocal
  Interventions: Device: Monofocal IOL

INTERVENTIONS:
Device: EDF — Extended depth of focus
  Arms: EDF
Device: Monofocal IOL — Monofocal
  Arms: Monofocal

SUMMARY:
EDF intraocular lens versus Monofocal intraocular lens

DETAILED DESCRIPTION:
Extended depth of Focus intraocular lens versus a monofocal intraocular lens

ELIGIBILITY:
Inclusion Criteria:

1. Patients of any gender, aged 18 years or older
2. Patient with clinically significant bilateral age-related cataracts planned for phacoemulsification cataract extraction and eligible for implantation of a posterior chamber intraocular lens as determined by investigator's medical judgement
3. Preoperative keratometric (corneal) astigmatism of 1.00 D or less (≤1.00 D)
4. Calculated lens power within the available range
5. Clear intraocular media other than cataract
6. Patient is willing and capable of providing informed consent
7. Patient is willing and capable of complying with visits and procedures as defined by this protocol

Exclusion Criteria:

1. Preoperative corrected distance visual acuity (CDVA) better than 0.3 logMAR (0.5 decimal)
2. Endothelial cell count of less than 2000/mm2
3. Acute, chronic, or uncontrolled systemic disease that could increase the operative risk or confound the outcome including but not limited to poorly controlled diabetes mellitus, active cancer treatment, mental illness, dementia, immunocompromised, connective tissue disease, clinically significant atopic disease, etc.
4. Ocular condition that may predispose patient to future complications, per investigator's medical judgement, including but not limited to severe dry eye, anterior segment pathology, uncontrolled glaucoma, that would result in a visual acuity of 0.2 logMAR or worse during the study
5. Clinically significant corneal abnormalities, including corneal dystrophy (epithelial, stromal or endothelial dystrophy), irregularity or oedema as per Investigator's medical judgement; conditions including but not limited to kerato-uveitis, keratopathy, keratectasia
6. Previous intraocular or corneal/refractive surgery that might confound the outcome of the investigation or increase the risk to the patient (including corneal transplants, removal of pterygium, and LASIK, LASEK, PRK, RK limbal relaxing incision etc.)
7. Any clinically significant condition that could affect IOL stability (e.g. zonular dialysis, evident zonular weakness or dehiscence, etc.)
8. Patients with diagnosed degenerative visual disorders (e.g. macular degeneration or other retinal disorders, optic nerve atrophy etc.) or any other pathologies of the eye that are predicted to result in a visual acuity of 0.2 logMAR or worse during the study
9. Current systemic or ocular pharmacotherapy that effects patients' vision with significant ocular side effects or any medications that could confound the outcome or increase subject risk
10. Clinically significant gonioscopic abnormalities
11. Amblyopia, strabismus, single eye status
12. Rubella, congenital, traumatic or complicated cataracts
13. History of or current anterior or posterior segment inflammation, including but not limited to iritis or uveitis
14. Microphthalmos or macrophthalmos
15. Pupil abnormalities (e.g. aniridia, abnormal shaped pupils, nonreactive pupils)
16. Pseudoexfoliation
17. Keratoconus or irregular astigmatism
18. Inability to measure keratometry or biometry (including but not limited to cataract density, etc.)
19. Pathologic miosis
20. Pregnant, plan to become pregnant, lactating during the course of the investigation, or another condition with associated fluctuation of hormones that could lead to refractive changes
21. Patients unable to meet the limitations of the protocol or likely of non-cooperation during the trial
22. Patients whose freedom is impaired by administrative or legal order
23. Concurrent participation in another clinical investigation in the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Mean monocular DCIVA at 66 cm | 6 Months
Mean monocular CDVA at 4 m | 6 Months
Mean monocular DCVA at 1 m (equal to -1 D defocus) | 6 Months
Mean monocular negative defocus range at the 0.20 logMAR compared to control | 6 Months
Proportion of eyes achieving monocular photopic CDVA 0.30 logMAR or better | 6 Months

SECONDARY OUTCOMES:
Patient Reported Outcome (PRO) | 6 Months
  Proportion of subjects who respond "I didn't wear glasses or contact lenses at all in the last 7 days" to question "How often did you wear glasses or contact lenses to see in the last 7 days?" from Patient Reported Outcome (PRO) survey

CONTACTS AND LOCATIONS:
Locations (14):
- Bulgaria (3):
  - Eye Hospital Zora, Sofia
  - Specialized Ophthalmological Hospital for Active Treatment, Sofia
  - Medical Center "Vereya", Stara Zagora
- Czechia (3):
  - Nemocnice Havlíčkův, Havlíčkův Brod
  - OFTEX ocni, Pardubice
  - Oční Centrum, Prague
- Romania (3):
  - Oculus Eye Clinic, Bucharest
  - Ofta Total Clinic, Sibiu
  - Medoptic Clinic, Suceava
- Spain (5):
  - Oftalvist, Alicante
  - Hospital Universitario Ramón y Cajal, Madrid
  - OMIQ Hospital Universitari, Sant Cugat del Vallès
  - University Hopital Complex of Santiago de Compostela, Santiago de Compostela
  - Oftalvist, Valencia